CLINICAL TRIAL: NCT00661167
Title: Phase II Study of ABI-007 by Tri-weekly Schedule for Patients With Unresectable or Recurrent Gastric Cancer Refractory to 5-FU Containing Regimen.
Brief Title: Phase II Study of ABI-007 for Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Taiho10041040
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): ABI-007
  Interventions: Drug: ABI-007

INTERVENTIONS:
Drug: ABI-007 — ABI-007 260 mg/m2, IV on day 1 of each 21 day cycle. Number of cycles: until progression or unacceptable toxicity develops.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of tri-weekly ABI-007 for recurrence or unresectable gastric cancer patients who have received one prior regimen containing fluoropyrimidine and developed disease progression or recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed gastric adenocarcinoma
* Received one prior regimen containing fluoropyrimidine analogs and developed disease progression or recurrence
* Age: 20 - 74
* At least one measurable lesion by RECIST criteria

Exclusion Criteria:

* History of Taxans use
* Patients with another active malignancy
* Pre-existing peripheral neuropathy of Grade 2, 3, or 4 (per CTCAE)
* Chronic treatment with steroids

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-04; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Overall response rate | During chemotherapy

SECONDARY OUTCOMES:
Safety | During chemotherapy
Progression-free survival | Until progression
Overall survival | Over a year form randomaization
Disease control rate | Duration chemoterapy

CONTACTS AND LOCATIONS:
Overall Officials: Nagahiro Saijo, MD, Study Chair — Kinki University Hospital
Locations (10):
- Japan (10):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Shikoku Cancer Center, Matsuyama, Ehime
  - National Kyusyu Cancer Center, Fukuoka, Fukuoka
  - Kitasato University East Hospital, Sagamihara, Kanagawa
  - Kochi Health Sciences Center, Kochi, Kochi
  - Saku Central Hospital Nagano Prefectural Federation of Agricultural Cooperatives for Health and Welfare, Saku, Nagano
  - Osaka Medical College Hospital, Takatsuki, Osaka
  - Saitama International medical center-comprehensive cancer center, Saitama Medical University, Hidaka, Saitama
  - Shizuoka Cancer Center, Sunto, Shizuoka
  - Kouseiren Takaoka Hospital, Takaoka, Toyama

REFERENCES:
- [Derived] Sasaki Y, Nishina T, Yasui H, Goto M, Muro K, Tsuji A, Koizumi W, Toh Y, Hara T, Miyata Y. Phase II trial of nanoparticle albumin-bound paclitaxel as second-line chemotherapy for unresectable or recurrent gastric cancer. Cancer Sci. 2014 Jul;105(7):812-7. doi: 10.1111/cas.12419. Epub 2014 Jul 7. PMID 24716542